CLINICAL TRIAL: NCT00308724
Title: Treating Late-Life Generalized Anxiety Disorder (GAD) in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Institutes of Health (NIH) (NIH); The University of Texas Health Science Center, Houston (Other); Kelsey Research Foundation (Other); Kelsey-Seybold Clinic (Other); Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Melinda Stanley, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H15958; R01MH053932 (NIH); NCT00081393 (obsolete NCT alias)
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; Geriatric
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Cognitive Behavior Therapy
  Interventions: Behavioral: Cognitive Behavior Therapy
- 2 (Active Comparator): Usual Care
  Interventions: Behavioral: Telephone check-in

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — 8 to 10 in person CBT sessions up to 60 minutes in duration within a 12 week time period
  Other Names: CBT
  Arms: 1
Behavioral: Telephone check-in — Biweekly telephone calls to monitor symptom severity, an enhanced Usual Care condition
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether cognitive behavior therapy (CBT) is effective in the treatment of generalized anxiety disorder (GAD) in adults age 60 and older in a primary care setting.

DETAILED DESCRIPTION:
Generalized Anxiety Disorder (GAD) is one of the most common anxiety disorders among older adults. Anxiety in older adults is associated with decreased physical activity, poorer self-perceptions of health, decreased life satisfaction, and increased loneliness. Because many older adults with anxiety seek assistance in a medical setting, treatment has been primarily pharmacological. There is, however, limited evidence of the effectiveness of psychotropic medications. Given the potential difficulties in prescribing psychotropic medications in later life (e.g., increased adverse effects, potential drug interactions), psychosocial treatments may be important alternative or adjuncts.

The treatment phase of this study lasts 10 weeks, during which patients will be randomly assigned to either cognitive behavior therapy (CBT) or usual care. Follow-up will last 12 months after treatment completion, during which time patients will complete telephone assessments.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Generalized Anxiety Disorder

Exclusion Criteria:

* Active suicidal intent
* Current psychosis
* Current bipolar disorder
* Substance abuse within past month
* Cognitive impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2004-03; Primary Completion 2008-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Anxiety | Baseline and 3, 6, 9, 12 and 15 months

SECONDARY OUTCOMES:
Functional and health status | Baseline and 3, 6, 9, 12 and 15 months
Quality of life inventory (QOLI) | Baseline and 3, 6, 9, 12 and 15 months
Satisfaction with CBT and general health care | Baseline and 3, 6, 9, 12 and 15 months
Service utilization | Baseline and 3, 6, 9, 12 and 15 months
Depression | Baseline and 3, 6, 9, 12 and 15 months
Sleep quality | Baseline and 3, 6, 9, 12 and 15 months
Use of alcohol and other substances | Baseline and 3, 6, 9, 12 and 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Melinda A. Stanley, Ph.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Houston Center for Quality of Care and Utilization Studies, Houston, Texas, United States

REFERENCES:
- [Background] Wetherell JL, Lenze EJ, Stanley MA. Evidence-based treatment of geriatric anxiety disorders. Psychiatr Clin North Am. 2005 Dec;28(4):871-96, ix. doi: 10.1016/j.psc.2005.09.006. No abstract available. PMID 16325733
- [Background] Stanley MA, Kunik ME. Anxiety in primary care: a frontier for mental health services research. Med Care. 2005 Dec;43(12):1161-3. doi: 10.1097/01.mlr.0000190923.04095.80. No abstract available. PMID 16299425
- [Background] Stanley MA, Hopko DR, Diefenbach GJ, Bourland SL, Rodriguez H, Wagener P. Cognitive-behavior therapy for late-life generalized anxiety disorder in primary care: preliminary findings. Am J Geriatr Psychiatry. 2003 Jan-Feb;11(1):92-6. PMID 12527544
- [Derived] Shrestha S, Stanley MA, Wilson NL, Cully JA, Kunik ME, Novy DM, Rhoades HM, Amspoker AB. Predictors of change in quality of life in older adults with generalized anxiety disorder. Int Psychogeriatr. 2015 Jul;27(7):1207-15. doi: 10.1017/S1041610214002567. Epub 2014 Dec 12. PMID 25497362
- [Derived] Stanley MA, Wilson NL, Novy DM, Rhoades HM, Wagener PD, Greisinger AJ, Cully JA, Kunik ME. Cognitive behavior therapy for generalized anxiety disorder among older adults in primary care: a randomized clinical trial. JAMA. 2009 Apr 8;301(14):1460-7. doi: 10.1001/jama.2009.458. PMID 19351943